CLINICAL TRIAL: NCT04662541
Title: Using Mobile Integrated Health and Telehealth to Support Transitions of Care Among Heart Failure Patients - Parent Study
Brief Title: Mobile Integrated Health in Heart Failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Ruth Masterson Creber, Professor of Nursing, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAU2716; IHS-2019C2-17373 (Other Grant/Funding Number: PCORI); 20-08022605-01 (Other: BRANY IRB while at WeillMC)
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
Keywords: Mobile Health; Mobile Integrated Health (MIH); Heart Failure (HF); mHealth
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Integrated Health (MIH) (Experimental): Patients with urgent medical needs are seen and treated in the home by trained community paramedics. The community paramedics perform a standardized assessment, including a physical examination, vital signs, home safety evaluation, and medication reconciliation. During the MIH encounter, the emergency medicine physician at each site is contacted via telemedicine. Physicians can access clinical notes, discharge summaries, and medication lists via the institutional EHR. Adjustments to outpatient medications can be e-prescribed and follow-up appointments can be scheduled with primary care clinicians.
  Interventions: Other: Mobile Integrated Health (MIH)
- Transitions of care coordinator (TOCC) (Active Comparator): Patients receive a follow-up phone calls for a nurse coordinator within 48-72 hours of hospital discharge. Phone calls include clinical/social needs assessment with escalation to primary care team, emergency care, or social work as needed; patient education; and reminder about follow-up appointments.
  Interventions: Other: Transitions of care coordinator (TOCC)

INTERVENTIONS:
Other: Mobile Integrated Health (MIH) — MIH leverages paramedics in the community and telemedicine (technology-enabled communication for health purposes) to provide medical care to heart failure patients in the home.
  Arms: Mobile Integrated Health (MIH)
Other: Transitions of care coordinator (TOCC) — The TOCC group will receive a follow-up phone call shortly after discharge in which the patient is assessed and connected to clinical and social services as needed and patient education is reinforced.
  Arms: Transitions of care coordinator (TOCC)

SUMMARY:
The purpose of this study is to compare how two different types of care after a hospitalization reduce hospital readmissions and symptom burden. The two types of care are a Transitions of Care Coordinator and Mobile Integrated Health. In the Transitions of Care Coordinator group, participants will receive a phone call from a care coordinator right after they go home following a hospitalization to check in. In the Mobile Integrated Health group, participants will be offered access to a community paramedic in case they need medical care while they are recovering at home after a hospitalization. The community paramedic will come to their home to perform an evaluation and set up a visit with an emergency physician via video conference. They may receive treatment at home or be transported to the emergency department. The investigators will be compare how well a Transitions of Care Coordinator and Mobile Integrated Health reduce readmissions to the hospital within 30 days of discharge and improve patient-reported health-related quality of life. The investigators hypothesize that participants in the Mobile Integrated Health group will have fewer readmissions to the hospital within 30 days of discharge and better health-related quality of life compared to participants in the Transitions of Care Coordinator group.

DETAILED DESCRIPTION:
High 30-day readmission rates among heart failure (HF) patients (25% nationally) inflict substantial burden on both health systems and patients. The majority of hospital readmissions occur in the first seven days following a hospitalization for HF and are driven by lack of improvement in persistent symptoms. While early, proactive follow-up after hospital discharge can improve health outcomes and patient-reported quality of life, barriers within health systems (lack of appointment availability, transportation, limited ability to deliver medical therapies in the home) have hampered efforts to provide comprehensive follow-up. Evidence suggests that Mobile Integrated Health (MIH), involving community paramedicine coupled with telemedicine, may be an effective intervention to reduce readmissions. The long-term goal of this research is to provide rigorous evidence of MIH with a diverse, representative sample. In this pragmatic randomized clinical trial the investigators will compare MIH to a Transitions of Care Coordinator (TOCC) intervention.

Specifically, the investigators aim to compare the effectiveness of MIH versus TOCC on healthcare utilization (aim 1), patient-reported outcomes (PROs; aim 2), and healthcare quality (aim 3). The investigators will also evaluate the factors that support the adoption, implementation, and maintenance from the perspective of multiple key stakeholders (aim 4). Participants in this RCT will be randomized 1:1 to either MIH (intervention) or TOCC (comparator). All participants will be enrolled and randomized during a hospitalization for HF. Participants in MIH will receive a follow-up phone call and access to community paramedics who provide a comprehensive assessment in the home, and specific medical therapies while consulting with an emergency room physician in real-time via telemedicine. Participants in TOCC will receive a follow-up phone call within 48-72 hours of discharge and connection to appropriate services (social work, care coordination, home care) as needed. Participants in both groups will complete PROs using a rigorously developed, visually enhanced mobile PRO reporting system.

The study population will include patients at NewYork-Presbyterian (NYP) and Mount Sinai health systems, which are part of the New York City-based INSIGHT PCORI-funded clinical research network. The targeted sample size across the two sites is 2,100 patients (1,050 per arm). This record is for the parent PCORI-funded trial evaluating MIH among HF patients. There is a separate sub-study being conducted locally at NYP which is described in another record.

ELIGIBILITY:
Inclusion Criteria:

* Medicare or Medicaid recipient
* Current diagnosis of HF
* Receiving inpatient care at NewYork Presbyterian or Mount Sinai Health Systems
* Live in NYC

Exclusion Criteria:

* Non-English, Spanish, Mandarin, or French speaking
* Diagnosis of dementia or psychosis
* Anticipated discharge to, or current residence in, skilled nursing facility or rehab center
* Anticipated discharge to, or currently receiving, hospice including home hospice
* Current candidate for and awaiting heart transplant
* Current left ventricular assist device (LVAD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2005 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of all-cause hospital readmissions | 30 days
  Number of readmissions to the hospital for any reason following a hospitalization
Patient-reported health-related quality of life score assessed using the KCCQ | 30 days
  Patient-reported health-related quality of life score assessed using the Kansas City Cardiomyopathy Questionnaire 23-item scale (KCCQ-23). KCCQ-23 scores range from 0 to 100, with lower scores (closer to 0) indicating worse symptoms and physical functioning, and higher scores (closer to 100) indicating better symptoms and physical functioning.

SECONDARY OUTCOMES:
Number of preventable emergency department visits | 30 days
  Number of emergency department visits following a hospitalization that are considered preventable according to a previously validated algorithm
Number of preventable emergency department visits | 60 days
  Number of emergency department visits following a hospitalization that are considered preventable according to a previously validated algorithm
Number of preventable emergency department visits | 90 days
  Number of emergency department visits following a hospitalization that are considered preventable according to a previously validated algorithm
Number of preventable emergency department visits | 6 months
  Number of emergency department visits following a hospitalization that are considered preventable according to a previously validated algorithm
Number of unplanned hospital readmissions | 30 days
  Number of readmissions to the hospital following a hospitalization that are considered unplanned according to a validated algorithm
Number of unplanned hospital readmissions | 60 days
  Number of readmissions to the hospital following a hospitalization that are considered unplanned according to a validated algorithm
Number of unplanned hospital readmissions | 90 days
  Number of readmissions to the hospital following a hospitalization that are considered unplanned according to a validated algorithm
Number of unplanned hospital readmissions | 6 months
  Number of readmissions to the hospital following a hospitalization that are considered unplanned according to a validated algorithm
Number of days at home | 30 days
  Number of days at home (alive and not in a hospital or other medical facility) following a hospitalization
Patient-reported symptoms and functioning score assessed using PROMIS-29 | 30 days
  Patient-reported symptoms and functioning score, measured using the Patient-Reported Outcomes Measurement Information System 29-item survey (PROMIS-29). PROMIS-29 domains are scored separately: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with participation in social roles, and pain interference. Each domain is scored using a standardized T-score ranging from approximately 20 to 80, with lower scores indicating less of the symptom (i.e., less fatigue), and higher scores indicating more of the symptom (i.e., more fatigue).
Patient-reported symptoms and functioning score assessed using PROMIS-29 | 60 days
  Patient-reported symptoms and functioning score, measured using the Patient-Reported Outcomes Measurement Information System 29-item survey (PROMIS-29). PROMIS-29 domains are scored separately: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with participation in social roles, and pain interference. Each domain is scored using a standardized T-score ranging from approximately 20 to 80, with lower scores indicating less of the symptom (i.e., less fatigue), and higher scores indicating more of the symptom (i.e., more fatigue).
Patient-reported symptoms and functioning score assessed using PROMIS-29 | 90 days
  Patient-reported symptoms and functioning score, measured using the Patient-Reported Outcomes Measurement Information System 29-item survey (PROMIS-29). PROMIS-29 domains are scored separately: physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with participation in social roles, and pain interference. Each domain is scored using a standardized T-score ranging from approximately 20 to 80, with lower scores indicating less of the symptom (i.e., less fatigue), and higher scores indicating more of the symptom (i.e., more fatigue).
Patient self-care score assessed using the SCHFI | 30 days
  Patient self-care score assessed using the Self-Care of Heart Failure Index (SCHFI). SCHFI standardized scores are reported separately for each domain: self-care maintenance, self-care monitoring, and self-care management. Scores range from 0 to 100, with lower scores (closer to 0) representing worse self-care and higher scores (closer to 100) representing better self-care.
Patient self-care score assessed using the SCHFI | 60 days
  Patient self-care score assessed using the Self-Care of Heart Failure Index (SCHFI). SCHFI standardized scores are reported separately for each domain: self-care maintenance, self-care monitoring, and self-care management. Scores range from 0 to 100, with lower scores (closer to 0) representing worse self-care and higher scores (closer to 100) representing better self-care.
Patient self-care score assessed using the SCHFI | 90 days
  Patient self-care score assessed using the Self-Care of Heart Failure Index (SCHFI). SCHFI standardized scores are reported separately for each domain: self-care maintenance, self-care monitoring, and self-care management. Scores range from 0 to 100, with lower scores (closer to 0) representing worse self-care and higher scores (closer to 100) representing better self-care.
Patient-reported health-related quality of life score assessed using the KCCQ | 60 days
  Patient-reported health-related quality of life score assessed using the Kansas City Cardiomyopathy Questionnaire 23-item scale (KCCQ-23). KCCQ-23 scores range from 0 to 100, with lower scores (closer to 0) indicating worse symptoms and physical functioning, and higher scores (closer to 100) indicating better symptoms and physical functioning.
Patient-reported health-related quality of life score assessed using the KCCQ | 90 days
  Patient-reported health-related quality of life score assessed using the Kansas City Cardiomyopathy Questionnaire 23-item scale (KCCQ-23). KCCQ-23 scores range from 0 to 100, with lower scores (closer to 0) indicating worse symptoms and physical functioning, and higher scores (closer to 100) indicating better symptoms and physical functioning.
Number of all-cause hospital readmissions | 60 days
  Number of readmissions to the hospital for any reason following a hospitalization
Number of all-cause hospital readmissions | 90 days
  Number of readmissions to the hospital for any reason following a hospitalization
Number of all-cause hospital readmissions | 6 months
  Number of readmissions to the hospital for any reason following a hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ruth M. Masterson Creber, PhD, MSc, RN, Principal Investigator — Columbia University; Leah Shafran Topaz, BPT, MSc, Study Director — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Mount Sinai Health System, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - New York Presbyterian/Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masterson Creber R, Daniels B, Reading Turchioe M, Shafran Topaz L, Zhao Y, Choi J, Ellison M, Merchant RC, Blutinger E, Goyal P, Yu J, Weiner MG, Sholle E, Ramasubbu K, Alishetti S, Axsom K, Slotwiner D, Rao M, Diaz I, Spertus JA, Sharma R, Kaushal R. Mobile Integrated Health vs a Transitions of Care Coordinator for Patients Discharged After Heart Failure: The Mighty-Heart Randomized Clinical Trial. JAMA Intern Med. 2025 Nov 1;185(11):1341-1348. doi: 10.1001/jamainternmed.2025.4483. PMID 40952734
- [Derived] Masterson Creber RM, Daniels B, Munjal K, Reading Turchioe M, Shafran Topaz L, Goytia C, Diaz I, Goyal P, Weiner M, Yu J, Khullar D, Slotwiner D, Ramasubbu K, Kaushal R. Using Mobile Integrated Health and telehealth to support transitions of care among patients with heart failure (MIGHTy-Heart): protocol for a pragmatic randomised controlled trial. BMJ Open. 2022 Mar 10;12(3):e054956. doi: 10.1136/bmjopen-2021-054956. PMID 35273051